CLINICAL TRIAL: NCT02630355
Title: Randomized Controlled Trial of Remote Ischaemic Preconditioning to Protect Against Dialysis Induced Cardiac Injury in Haemodialysis: Low Vs. High Intensity
Brief Title: Remote Ischaemic Preconditioning to Prevent Dialysis Induced Cardiac Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely after ad-interim analysis for the primary outcome.
Sponsor: Western University, Canada (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Principal Investigator, Christopher McIntyre, Dr., Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-15-091
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Hemodialysis; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Sham Comparator): Inflation of blood pressure cuff in lower limb to 40mmHg for four cycles of 5 minutes inflation and then deflation
  Interventions: Other: Remote Ischaemic Preconditioning
- Low Intensity (Active Comparator): Inflation of blood pressure cuff in lower limb to 200mmHg for two cycles of 5 minute inflation and then deflation.
  Interventions: Other: Remote Ischaemic Preconditioning
- Standard Intensity (Active Comparator): Inflation of blood pressure cuff in lower limb to 200mmHg for four cycles of 5 minute inflation and then deflation.
  Interventions: Other: Remote Ischaemic Preconditioning
- High Intensity (Active Comparator): Inflation of blood pressure cuff in lower limb to 200mmHg for four cycles of 5 minute inflation and deflation on weekly basis for four consecutive weeks.
  Interventions: Other: Remote Ischaemic Preconditioning

INTERVENTIONS:
Other: Remote Ischaemic Preconditioning — Inflation of blood pressure cuff in lower limb

SUMMARY:
This study evaluates the use of remote ischaemic preconditioning for the prevention of dialysis induced cardiac injury. The study uses four arms to test different frequencies of application to ascertain which, if any, is most successful at reducing dialysis induced cardiac injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having haemodialysis treatment at least 3 times per week at a London Health Sciences Centre facility
2. Male and female, age≥16 years old.

Exclusion Criteria:

1. Not meeting inclusion criteria
2. Exposure to haemodialysis for <90 days prior to recruitment
3. Severe heart failure (New York Heart Association grade IV)
4. Cardiac transplant recipients
5. Mental incapacity to consent
6. Declined to participate
7. Taking cyclosporin
8. Taking ATP-sensitive potassium channel opening or blocking drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a reduction in the number of left ventricular segments undergoing a greater than 30% reduction in longitudinal strain as detected by echocardiography at final study visit | 4 weeks

SECONDARY OUTCOMES:
Number of segments undergoing >30% reduction in longitudinal strain at intervention, week 1, week 2 and week 3 visits | up to 3 weeks
Difference between pre and peak global longitudinal strain at intervention, week 1, week 2 and week 3 visits | up to 3 weeks
Change in pre-dialysis global longitudinal strain between baseline and final study visit | between 1 and 4 weeks
Change in Troponin-T, Plasma IL-6 and N-Type proBNP at intervention, first follow-up and final visit | up to 4 weeks

IPD SHARING:
Plan to Share IPD: No